CLINICAL TRIAL: NCT02196350
Title: The Impact of the P4 Approach, Preventive, Predictive, Personalized and Participatory in Newly Diagnosed Type 2 Diabetics in Hillegom
Brief Title: P4 Approach in Diabetes Type 2
Acronym: P4P-Hillegom
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: W.J. Pasman (Other)
Responsible Party: Sponsor-Investigator, W.J. Pasman, PhD, TNO
Organization: TNO (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: P9607
Record Dates: First submitted 2014-07-16; First posted 2014-07-22 (Estimated); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Type 2 Diabetes
Keywords: personalized treatment; prevention; improved diagnosis
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Intervention A: Diet (Experimental): Intervention A: One week of very low calorie diet, 12 weeks of low calorie diet; exercise according to the Dutch Norm for Healthy Behaviour (Nederlandse Norm Gezond Bewegen).
  Interventions: Behavioral: Intervention A: Diet
- Intervention B: Exercise (Experimental): Intervention B: Combination of strength and endurance training, 3 x per week 60 minutes according to the Exercise Program Diabetes (Beweegprogramma Diabetes).
  Healthy isocaloric diet.
  Interventions: Behavioral: Intervention B: Exercise
- Intervention C: Diet and Exercise (Experimental): Intervention C: one week very low calorie diet, followed by 12 weeks healthy isocaloric diet.
  One week exercise according to the Dutch Norm for Healthy Behaviour (Nederlandse Norm Gezond Bewegen) followed by 12 weeks strength and endurance training (3 x per week 60 minutes) according to the Exercise Program Diabetes (Beweegprogramma Diabetes)
  Interventions: Behavioral: Intervention C: Diet and Exercise
- Control - Historical data (No Intervention): Historical data from the GPs Information System from 60 newly diagnosed type 2 diabetes patients in the last five years will be used as control.

INTERVENTIONS:
Behavioral: Intervention A: Diet — subjects visit the dietitian at week 0, 1, 2, 6, 10 and 13 for dietary advice
  Other Names: very low calorie diet based on Modifast meal replacers.
  Arms: Intervention A: Diet
Behavioral: Intervention B: Exercise — subjects visit the physiotherapist three times weekly; subjects visit the dietitian at week 0, 1, 2, 6, 10 and 13 for dietary advice.
  Arms: Intervention B: Exercise
Behavioral: Intervention C: Diet and Exercise — subjects visit the physiotherapist three times weekly; subjects visit the dietitian at week 0, 1, 2, 6, 10 and 13 for dietary advice.
  Other Names: very low calorie diet based on Modifast meal replacers.
  Arms: Intervention C: Diet and Exercise

SUMMARY:
The study aims to assess the impact of the P4 approach on established markers of glucose metabolism in type 2 diabetics.

Secondary objectives are examination of the changes in physical characteristics, quality of life and the indices for beta cell function, hepatic insulin resistance and muscle insulin resistance .

DETAILED DESCRIPTION:
This study will be a proof-of-principle exploratory study. Subjects in the P4 program will receive a personalized diagnosis and treatment. After investigation of the status of the different organs involved in diabetes (liver, muscle, pancreas), subjects in the P4 group are divided into 3 subgroups. Each subgroup receives a personalized lifestyle advice. This lifestyle advice may comprise different interventions, i.e. very low calorie diet, low calorie diet, strength training, endurance training. Dependent on the type of intervention, these interventions will be supervised by a dietitian or physiotherapist.

All subjects will visit a central study center 5 times during the study and 3 times during follow-up. During these visits physical measures will be taken and data will be collected by the general practitioner assistant.

After the three month intervention period the subjects will return to usual care via the general practitioner.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy as assessed by the

   * health and lifestyle questionnaire, (P9607 F02; in Dutch)
   * physical examination
   * results of the pre-study laboratory tests
2. Age 30-80 years
3. Stable BMI 25-35 kg/m2
4. Diagnosis diabetes type 2 based upon:

   Fasting glucose >6.9 mmol/l on two different days or one measurement of non-fasting glucose >11.0 mmol/l in combination with symptoms of hyperglycemia
5. Duration of diabetes maximally 1 year
6. Informed consent signed;
7. Willing to comply with the study procedures during the study;
8. Appropriate veins for blood sampling/ cannula insertion according to the general practitioner assistant (GPA);
9. Voluntary participation
10. Physically able to perform training activities
11. Willing to accept use of all nameless data, including publication, and the confidential use and storage of all data for at least 15 years.

Exclusion Criteria:

1. Use of insulin, corticosteroids (systemic), or beta-blockers in past month
2. Diabetes occurring after several attacks of pancreatitis known as pancreatic diabetes
3. Slow onset type 1 diabetes
4. Use of oral diabetes medication in past year
5. (Having a history of a) medical condition that might significantly affect the study outcome as judged by the medical investigator and health and life style questionnaire. This includes diabetes type 1, gastrointestinal dysfunction, diseases related to inflammation or allergy, or a psychiatric disorder.
6. Hypertension: systolic blood pressure >160 mmHg, diastolic blood pressure >90 mmHg
7. Kidney problems based upon proteinuria and creatinine >150 mmol/l
8. Insufficient beta cell function based on Disposition index < 1.5 as determined during the OGTT in study on day 01*
9. Physical activity higher than according to the Diabetes guidelines (moderate intensity one hour a day, seven days a week (overweight adults))
10. Alcohol consumption > 21 (women) - 28 (men) units/week
11. Reported unexplained weight loss or gain of > 2 kg in the month prior to the pre-study screening
12. Recent blood donation (<1 month prior to the start of the study)
13. Not willing to give up blood donation during the study
14. Personnel of TNO and their partner
15. Not having a general practitioner
16. Not willing to accept information-transfer concerning participation in the study, or information regarding his health, like laboratory results, findings at anamnesis or physical examination and eventual adverse events to and from his general practitioner.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c levels | In-study at week 0 (baseline) and 13 (end of study); follow-up after 6, 12 and 24 months
  Changes in primary outcome measures will be determined by using a mixed model
Change in 2h glucose levels | In-study at week 0 (baseline) and 13;
  2h glucose will be measured after Oral Glucose Tolerance Test (OGTT). Changes in primary outcome measures will be determined by using a mixed model
Change in fasting blood glucose levels | In-study at week 0 (baseline) and 13 (end of study); follow-up after 6, 12 and 24 months
  After 8 hour fasting. Changes in primary outcome measures will be determined by using a mixed model.
percentage of participants that reach normoglycemia | end of study (after 13 weeks)
  normoglycemia is determined by fasting blood glucose level of less than 6.1 mmol/L

SECONDARY OUTCOMES:
body weight | screening; in-study at week 0, 4, 8 and 13; during follow up after 6, 12 and 24 months
  measured by the general practitioner assistant
blood pressure | screening; in-study at week 0, 4, 8 and 13; during follow up after 6, 12 and 24 months
  measured by the general practitioner assistant
waist circumference | screening; in-study at week 0, 4, 8 and 13; during follow up after 6, 12 and 24 months
  measured by general practitioner assistant
body fat percentage | screening; in-study at week 0, 4, 8 and 13; during follow up after 6, 12 and 24 months
  measured by general practitioner assistant
change indices for muscle insulin resistance | screening; in-study at week 0 and 13;
  at week 0 and 13 the indices will be calculated from Oral glucose tolerance test data.
  Blood will be collected at the blood collection centre in Hillegom
health behaviour change | in-study at week 0, 13; during follow-up at 6, 12 and 24 months
  established by comparing baseline values with end of study values for food intake and physical activity as measured by a Lifestyle-questionnaire
change in vitality as assessed with a vitality questionnaire (Vita-16) | in-study at week 0, 13; during follow-up at 6, 12 and 24 months
change in subjective quality of life as assessed with RAND-36 questionnaire | in-study at week 0, 13; during follow-up at 6, 12 and 24 months
change in indices for beta cell function | screening; in-study at week 0 and 13;
  at week 0 and 13 the indices will be calculated from Oral glucose tolerance test data.
  Blood will be collected at the blood collection centre in Hillegom
change in indices for hepatic insulin resistance | screening; in-study at week 0 and 13;
  at week 0 and 13 the indices will be calculated from Oral glucose tolerance test data.
  Blood will be collected at the blood collection centre in Hillegom

CONTACTS AND LOCATIONS:
Overall Officials: Wilrike Pasman, PhD, Principal Investigator — Netherlands Organisation for Applied Scientific Research (TNO); Peter van Dijken, Dr., Study Director — Netherlands Organisation for Applied Scientific Research (TNO)
Locations (9):
- Netherlands (9):
  - Huisartsenpraktijk Lommelaars, Hillegom, South Holland
  - Huisartspraktijk C.C. Dekker, Hillegom, South Holland
  - Huisartspraktijk Tubbergen, Hillegom, South Holland
  - Huisartsenpraktijk Sixlaan 9, Hillegom, South Holland
  - Huisartsenpraktijk J.G. van Dusseldorp, Hillegom, South Holland
  - Huisartsenpraktijk van der Kaaden, Hillegom, South Holland
  - Huisartsenpraktijk Elsbroek, Hillegom, South Holland
  - Huisartsenpraktijk Mulders, Hillegom, South Holland
  - Netherlands Organisation for Applied Scientific Research (TNO), Zeist, Utrecht